CLINICAL TRIAL: NCT02624960
Title: Safety and Performance of the AccuCinch® Ventricular Repair System
Brief Title: Safety and Performance of the AccuCinch® System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew and updated study design. Refer to NCT03183895.
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4432
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure; Mitral Valve Insufficiency
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accucinch Implant (Experimental): Accucinch Implant procedure is completed
  Interventions: Device: Accucinch Implant

INTERVENTIONS:
Device: Accucinch Implant — Percutaneous implantation of the Accucinch Implant in the mitral subannular space

SUMMARY:
This is a single-arm, multi-center, open-label controlled study that will assess the safety and performance of the Accucinch System to induce left ventricular reverse remodeling and reduce the severity of functional mitral regurgitation in symptomatic adult patients with mitral regurgitation and left ventricular remodeling due to dilated cardiomyopathy (ischemic or non-ischemic etiology), who are of high operative risk.

ELIGIBILITY:
Inclusion Criteria:

* Study patient is an adult of legal consent age
* Severity of FMR: ≥ Moderate
* Ejection Fraction: ≥20 to ≤60%
* Symptom Status: NYHA II-IVa
* Treatment and compliance with optimal guideline directed medical therapy for heart failure for at least 1 month
* Surgical risk: Subject is eligible for cardiac surgery

Exclusion Criteria:

* Patients with significant organic mitral valve pathology (e.g. myxomatous degeneration, mitral valve prolapse or flail leaflets)
* Myocardial infarction or any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
* Prior surgical, transcatheter, or percutaneous mitral valve intervention
* Untreated clinically significant coronary artery disease requiring revascularization
* Hemodynamic instability: Hypotension or requirement for inotropic support or mechanical hemodynamic support
* Any planned cardiac surgery or interventions within the next 6 months
* NYHA class IVb (i.e., non-ambulatory) or ACC/AHA Stage D heart failure
* Fixed pulmonary artery systolic pressure >70 mmHg
* Severe tricuspid regurgitation
* Modified Rankin Scale ≥ 4 disability
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
* Mitral valve area less than 4.0 cm2
* Anatomical pathology/constraints preventing appropriate access/implant of the GDS Accucinch System
* Renal insufficiency
* Mitral annular calcification
* Moderate or severe aortic valve stenosis or regurgitation or aortic valve prosthesis
* Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus or vegetation
* Active bacterial endocarditis
* History of stroke within the prior 3 months
* Subjects in whom anticoagulation is contraindicated
* Anemia
* Thrombocytopenia or thrombocytosis
* Bleeding disorders or hypercoaguable state
* Active peptic ulcer or active gastrointestinal bleeding
* Known allergy to nitinol, polyester, or polyethylene
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure.
* Life expectancy < 1 year due to non-cardiac conditions
* Currently participating in another interventional investigational study
* Implant or revision of any rhythm management device or implantable cardioverter defibrillator within the prior month
* Absence of CRT with class I indication criteria for biventricular pacing - Subjects on high dose steroids or immunosuppressant therapy
* Female subjects who are pregnant, of child bearing potential or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The additive reduction in the mitral annular axial dimensions (anteroposterior plus commissure-to-commissure axes) measured via echocardiography, paired by subject | 6 months
  The differences between baseline and 6 months in the sum of the two annulus measures will be calculated for each subject and the mean change tested via the paired t-test.

SECONDARY OUTCOMES:
Device Success: Percentage of patients in whom all pre-specified device performance endpoints are met but no pre-specified device complications are met. | 30 Days, 6 months, 12 months, and 2 years
  Pre-specified endpoints are the following:stroke-free survival AND intended positioning of the original implant AND No additional surgical or interventional procedures AND intended performance of the device (no migration, embolization, fracture, thrombosis, etc AND reduction of MR by at least one grade and reduction of combined mitral annular diameters by at least 20%) AND no device-related complications (erosion, migration, etc.) at 30-days and all subsequent follow-up time points.
Procedural Safety: Incidence rate of the occurrence of the individual pre-specified safety events that occur within 30 days of the index procedure | 30 days after the index procedure
  Pre-specified safety events include the following:
  * Death
  * Stroke
  * Life-threatening or Extensive bleeding (MVARC scale)
  * Major vascular complications
  * Major cardiac access (e.g., structural) complications
  * Stage 2 or 3 acute kidney injury (AKI)
  * New myocardial infarction or coronary insufficiency requiring PCI or CABG
  * Severe hypotension, heart failure, or respiratory failure
  * Any implant-related dysfunction or other complication requiring surgery or unplanned intervention or prolonged intubation > 24 hours
Long Term Safety: Incidence rate of the occurrence of the individual pre-specified safety events at 6 months, 1 year, and 2 years. | 6 months, 1 year, 2 years post index procedure
  Pre-specified endpoints include the following:
  * Death, cardiac, non-cardiac
  * Stroke
  * Mitral valve reintervention or surgery
  * MI
  * Any device related complication/ dysfunction
  * New atrial fibrillation (AF)
  * New conduction disturbance requiring permanent pacemaker (PM)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schofer, MD, PhD, Principal Investigator — Medical Director, Medical Care Center Hamburg; Dept Chief, Percutaneous Treatment of Structural Heart Disease, Albertinen Heart Center, Hamburg Germany

IPD SHARING:
Plan to Share IPD: No